CLINICAL TRIAL: NCT05082402
Title: Imaging of Retinochoroidal Vasculature in Patients Being Assessed for Cardiovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rukhsana Mirza, Principal Investigator, M.D., MS, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00215189
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Retina; Change
Keywords: retinal vasculature; cardiovascular disease; swept source optical coherence tomography angiography; SS-OCTA; carotid duplex ultrasonography
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All Participants (Experimental): 50 participants identified in the Northwestern Medicine Division of Vascular Surgery.
  Interventions: Diagnostic Test: Swept Source Optical Coherence Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Swept Source Optical Coherence Tomography Angiography — The PLEX Elite 9000 is an FDA cleared research device for use in ocular imaging obtained by Northwestern University by way of a purchase agreement with the manufacturer, Carl Zeiss Meditec, Inc. It is currently unavailable outside of participation in the ARI Network, a cloudbased storage and image processing platform using deidentified information shared between academic institutions. The ARI Network is managed by a group of physicians and scientists from around the world that are working to better understand eye diseases.

SUMMARY:
This study aims to determine whether changes in retinal vasculature seen on SS-OCTA can be correlated to degree of cardiovascular disease as measured by carotid duplex ultrasonography.

DETAILED DESCRIPTION:
The study's primary objective is to determine whether measures taken from SS-OCTA, color fundus photography, and retinal exams can correlate with and predict the presence/degree of carotid occlusive disease as determined by carotid duplex ultrasonography by examining the following parameters: retinal vessel caliber, retinal vessel density, retinal vessel perfusion, retinal vessel tortuosity, presence of Hollenhorst or other plaques, and/or areas of ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 80 years of age.
* No known prior history of retinal disease.
* Able to participate in a clinical eye examination setting.
* Able to consent.
* Subjects receiving standard of care carotid duplex ultrasounds.

Exclusion Criteria:

* Known ophthalmologic disease (e.g. glaucoma, macular degeneration, ocular injury) other than corrected refractive error.
* Lack of capacity to provide informed consent.
* Subjects younger than 18 years of age or older than 80 years of age.
* History of stroke or acute loss of vision.
* Unable to participate in a clinical eye examination setting.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation with and prediction of the presence/degree of carotid occlusive disease as determined by carotid duplex ultrasonography | 2 hours
  Determining whether measures taken from SS-OCTA, color fundus photography, and retinal exams can correlate with and predict the presence/degree of carotid occlusive disease as determined by carotid duplex ultrasonography by examining the following parameters: retinal vessel caliber, retinal vessel density, retinal vessel perfusion, retinal vessel tortuosity, presence of Hellenhorst or other plaques, and/or areas of ischemia.

CONTACTS AND LOCATIONS:
Overall Officials: Rukhsana Mirza, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University/Northwestern Medical Group, Department of Ophthalmology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Climie RE, van Sloten TT, Bruno RM, Taddei S, Empana JP, Stehouwer CDA, Sharman JE, Boutouyrie P, Laurent S. Macrovasculature and Microvasculature at the Crossroads Between Type 2 Diabetes Mellitus and Hypertension. Hypertension. 2019 Jun;73(6):1138-1149. doi: 10.1161/HYPERTENSIONAHA.118.11769. No abstract available. PMID 31067192
- [Background] Cade WT. Diabetes-related microvascular and macrovascular diseases in the physical therapy setting. Phys Ther. 2008 Nov;88(11):1322-35. doi: 10.2522/ptj.20080008. Epub 2008 Sep 18. PMID 18801863
- [Background] Wang SB, Mitchell P, Plant AJ, Phan K, Liew G, Thiagalingam A, Burlutsky G, Gopinath B. Metabolic syndrome and retinal microvascular calibre in a high cardiovascular disease risk cohort. Br J Ophthalmol. 2016 Aug;100(8):1041-6. doi: 10.1136/bjophthalmol-2015-307637. Epub 2015 Nov 3. PMID 26531050
- [Background] Zhao Y, Yang K, Wang F, Liang Y, Peng Y, Shen R, Wong T, Wang N. Associations between metabolic syndrome and syndrome components and retinal microvascular signs in a rural Chinese population: the Handan Eye Study. Graefes Arch Clin Exp Ophthalmol. 2012 Dec;250(12):1755-63. doi: 10.1007/s00417-012-2109-2. Epub 2012 Sep 5. PMID 22948948
- [Background] Michelson EL, Morganroth J, Nichols CW, MacVaugh H 3rd. Retinal arteriolar changes as an indicator of coronary artery disease. Arch Intern Med. 1979 Oct;139(10):1139-41. PMID 485746
- [Background] Phan K, Mitchell P, Liew G, Plant AJ, Wang SB, Au C, Chiha J, Kovoor P, Thiagalingam A, Burlutsky G, Gopinath B. Association between Retinal Arteriolar and Venule Calibre with Prevalent Heart Failure: A Cross-Sectional Study. PLoS One. 2015 Dec 11;10(12):e0144850. doi: 10.1371/journal.pone.0144850. eCollection 2015. PMID 26659133
- [Background] Wong TY, Cheung N, Islam FM, Klein R, Criqui MH, Cotch MF, Carr JJ, Klein BE, Sharrett AR. Relation of retinopathy to coronary artery calcification: the multi-ethnic study of atherosclerosis. Am J Epidemiol. 2008 Jan 1;167(1):51-8. doi: 10.1093/aje/kwm256. Epub 2007 Sep 24. PMID 17893402
- [Background] Liew G, Mitchell P, Chiha J, Plant AJH, White A, Joachim N, Wang S, Burlutsky G, Kovoor P, Thiagalingam A, Gopinath B. Retinal microvascular changes in microvascular angina: Findings from the Australian Heart Eye Study. Microcirculation. 2019 Aug;26(6):e12536. doi: 10.1111/micc.12536. Epub 2019 Mar 20. PMID 30758094
- [Background] Liew G, Wang JJ, Mitchell P, Wong TY. Retinal vascular imaging: a new tool in microvascular disease research. Circ Cardiovasc Imaging. 2008 Sep;1(2):156-61. doi: 10.1161/CIRCIMAGING.108.784876. PMID 19808533
- [Background] Tabatabaee A, Asharin MR, Dehghan MH, Pourbehi MR, Nasiri-Ahmadabadi M, Assadi M. Retinal vessel abnormalities predict coronary artery diseases. Perfusion. 2013 May;28(3):232-7. doi: 10.1177/0267659112473173. Epub 2013 Jan 15. PMID 23322671
- [Background] Wang SB, Mitchell P, Liew G, Wong TY, Phan K, Thiagalingam A, Joachim N, Burlutsky G, Gopinath B. A spectrum of retinal vasculature measures and coronary artery disease. Atherosclerosis. 2018 Jan;268:215-224. doi: 10.1016/j.atherosclerosis.2017.10.008. Epub 2017 Oct 10. PMID 29050745
- [Background] Cheung N, Bluemke DA, Klein R, Sharrett AR, Islam FM, Cotch MF, Klein BE, Criqui MH, Wong TY. Retinal arteriolar narrowing and left ventricular remodeling: the multi-ethnic study of atherosclerosis. J Am Coll Cardiol. 2007 Jul 3;50(1):48-55. doi: 10.1016/j.jacc.2007.03.029. Epub 2007 Jun 18. PMID 17601545
- [Background] Wang L, Wong TY, Sharrett AR, Klein R, Folsom AR, Jerosch-Herold M. Relationship between retinal arteriolar narrowing and myocardial perfusion: multi-ethnic study of atherosclerosis. Hypertension. 2008 Jan;51(1):119-26. doi: 10.1161/HYPERTENSIONAHA.107.098343. Epub 2007 Nov 12. PMID 17998474
- [Background] Murray CSG, Nahar T, Kalashyan H, Becher H, Nanda NC. Ultrasound assessment of carotid arteries: Current concepts, methodologies, diagnostic criteria, and technological advancements. Echocardiography. 2018 Dec;35(12):2079-2091. doi: 10.1111/echo.14197. PMID 30506607
- [Background] Kadian-Dodov D, Papolos A, Olin JW. Diagnostic utility of carotid artery duplex ultrasonography in the evaluation of syncope: a good test ordered for the wrong reason. Eur Heart J Cardiovasc Imaging. 2015 Jun;16(6):621-5. doi: 10.1093/ehjci/jeu315. Epub 2015 Feb 10. PMID 25669837
- [Background] Lahme L, Marchiori E, Panuccio G, Nelis P, Schubert F, Mihailovic N, Torsello G, Eter N, Alnawaiseh M. Changes in retinal flow density measured by optical coherence tomography angiography in patients with carotid artery stenosis after carotid endarterectomy. Sci Rep. 2018 Nov 21;8(1):17161. doi: 10.1038/s41598-018-35556-4. PMID 30464189
- [Background] Wong TY, Klein R, Klein BE, Tielsch JM, Hubbard L, Nieto FJ. Retinal microvascular abnormalities and their relationship with hypertension, cardiovascular disease, and mortality. Surv Ophthalmol. 2001 Jul-Aug;46(1):59-80. doi: 10.1016/s0039-6257(01)00234-x. PMID 11525792
- [Background] Heitmar R, Cubbidge RP, Lip GY, Gherghel D, Blann AD. Altered blood vessel responses in the eye and finger in coronary artery disease. Invest Ophthalmol Vis Sci. 2011 Aug 3;52(9):6199-205. doi: 10.1167/iovs.10-6628. PMID 21474768
- [Background] McClintic BR, McClintic JI, Bisognano JD, Block RC. The relationship between retinal microvascular abnormalities and coronary heart disease: a review. Am J Med. 2010 Apr;123(4):374.e1-7. doi: 10.1016/j.amjmed.2009.05.030. PMID 20362758
- [Background] Wang J, Jiang J, Zhang Y, Qian YW, Zhang JF, Wang ZL. Retinal and choroidal vascular changes in coronary heart disease: an optical coherence tomography angiography study. Biomed Opt Express. 2019 Mar 4;10(4):1532-1544. doi: 10.1364/BOE.10.001532. eCollection 2019 Apr 1. PMID 31061756